CLINICAL TRIAL: NCT01738685
Title: Intervention to Improve Self-Care of Symptoms in Breast Cancer Survivors on Adjuvant Endocrine Therapy.
Acronym: Relief
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Van Londen, Gijsberta, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO12050094
Record Dates: First submitted 2012-11-15; First posted 2012-11-30 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer.; Adjuvant Endocrine therapy.
MeSH Terms: conditions — Breast Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control. (Other): Nutritional Education.
  Interventions: Other: Nutritional Education.
- Behavioral Intervention (Other): Behavioral Intervention.
  Interventions: Behavioral: Behavioral Intervention.

INTERVENTIONS:
Behavioral: Behavioral Intervention.
  Arms: Behavioral Intervention
Other: Nutritional Education.
  Arms: Control.

SUMMARY:
Hormone responsive breast cancer is common and costly. Long-term adjuvant endocrine therapy (AET) improves breast cancer outcomes greatly, but, unfortunately, is commonly associated with physical and emotional concerns. I propose to evaluate the feasibility and preliminary effectiveness of a behavioral intervention to facilitate problem identification, provide education, coaching for breast cancer survivors with symptoms while on AET. Therefore, the intervention intends to empower women to engage in better self-care and seek out resources they need, which, in turn, will lead to better symptom management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50.
* Nonmetastatic bread cancer survivors reporting being bothered by 1 or more symptoms related to their treatment with AET (for > 0 months and < 6 months).
* Possess a household or cell telephone.
* Ability to provide informed consent.

Exclusion Criteria:

* Clinically significant cognitive impairment.
* Communication barrier limiting ability to participate in telephone assessments.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction determined by the Client Satisfaction Survey | Up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: G van Londen, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States